CLINICAL TRIAL: NCT06060327
Title: The Efficacy and Safety of Tranexamic Acid Versus Uterotonic Agents in Reducing Blood Loss During and After Cesarean Section Among High-risk Patients: a Comparative Study
Brief Title: Comparing Tranexamic Acid Versus Ecbolics in Preventing Hemorrhage During and After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-147-2021
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Postpartum Hemorrhage; Blood Loss, Postoperative; Cesarean Section Complications
MeSH Terms: conditions — Postpartum Hemorrhage; Postoperative Hemorrhage | interventions — Tranexamic Acid; Misoprostol; carbetocin; Oxytocin

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial including 4 groups comprising of 111 each.
  Group 1 will receive Oxytocin only, Group 2 will receive Oxytocin and Tranexamic acid, Group 3 will receive Oxytocin and Misoprostol and Group 4 will receive Oxytocin and Carbetocin.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oxytocin Group (Active Comparator): o In Oxytocin group (n=111), patients will receive 10 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) given as infusion in 500 ml lactated ringer/s solution at a rate of 125ml/hour after delivery of the placenta.
  Interventions: Drug: Tranexamic acid
- Tranexamic acid (Active Comparator): o In Tranexamic group (n=111), patients will be given 1 gm (10 ml) TXA (Kapron, Amoun, Egypt) diluted in 20 ml of Glucose 5% (administered as intravenous infusion over 5 minutes, at least 15 minutes prior to skin incision).
  Oxytocin 5 IU will be given slowly intravenous following delivery of the baby.
  Interventions: Drug: Tranexamic acid
- Misoprostol (Active Comparator): o In Misoprostol group (n=111), 400 microgram misoprostol (2 tablets - Cytotec, Pfizer, G.D. Searle LLC) will be inserted intraoperative inside the uterus after delivery of the placenta Oxytocin 5 IU will be given slowly intravenous following delivery of the baby.
  Interventions: Drug: Tranexamic acid
- Carbetocin (Active Comparator): o In carbetocin group (n=111) 100 microgram carbetocin (Pabal, Ferring, Kiel, Germany) will be given as an intravenous bolus dose following the delivery of the placenta.
  Oxytocin 5 IU will be given slowly intravenous following delivery of the baby.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Giving oxytocin only, or oxytocin in addition to Tranexamic acid, Misoprostol or Carbetocin the mentioned doses and by the mention routes, then comparing the estimated blood loss in each group.
  Other Names: Misoprostol; Carbetocin; Oxytocin

SUMMARY:
The study will include 444 pregnant patients undergoing cesarean section in Kasr Al Aini.

Following a proper medical history taking, examination will be done, investigations including laboratory tests and obstetric ultrasound will be done.

Then, the patients will be divided into 4 groups, receiving Oxytocin only (Group 1), Oxytocin + Tranexamic acid (Group 2), Oxytocin and Misoprostol (Group 3) or Oxytocin and Carbetocin (Group 4) followed by collection of necessary data.

DETAILED DESCRIPTION:
The study will include (444) pregnant women attending for cesarean delivery in Kasr El Aini hospital (faculty of medicine - Cairo university).

The following will be done to all participants:

* Informed written consent: after discussing the nature of the study as well as the expected value, outcome, and possible adverse effects.
* Full medical history: including full obstetric history and current pregnancy history (entailing the 1st day of LMP).
* Thorough Clinical Examination: general (maternal body weight and vital signs) and full obstetric examination.
* Obstetric ultrasonography: to confirm singleton pregnancy, gestational age and the eligibility of the current pregnancy to participate in the study.
* Preoperative laboratory tests: including prothrombin time, prothrombin concentration, complete blood count, and liver and kidney function tests.
* Group allocation: Before surgery, participants will be randomly and equally assigned into four groups; Tranexamic Acid group, Misoprostol group, Carbetocin group and Oxytocin group. Randomization will be performed using computer-generated random numbers.
* In Oxytocin group (n=111), patients will receive 10 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) given as infusion in 500 ml lactated ringer/s solution at a rate of 125ml/hour after delivery of the placenta.
* In Tranexamic group (n=111), patients will be given 1 gm (10 ml) TXA (Kapron, Amoun, Egypt) diluted in 20 ml of Glucose 5% (administered as intravenous infusion over 5 minutes, at least 15 minutes prior to skin incision).
* In Misoprostol group (n=111), 400 microgram misoprostol (2 tablets - Cytotec, Pfizer, G.D. Searle LLC) will be inserted intraoperative inside the uterus after delivery of the placenta.
* In carbetocin group (n=111) 100 microgram carbetocin (Pabal, Ferring, Kiel, Germany) will be given as an intravenous bolus dose following the delivery of the placenta.
* In all groups, patients will additionally receive 5 IU oxytocin given as slow intravenous bolus following delivery of the baby.
* All cesarean sections will be done under spinal anesthesia by the following operative steps: pfannenstiel incision, transverse lower uterine segment incision, immediate cord clamping (< 30 seconds) and the placenta will be removed by controlled cord traction after its spontaneous separation, closure of uterus in 2 layers, closure of anterior abdominal wall in anatomical manner (adequate hemostasis will be ensured in all operative steps).
* The number and the difference of weight of operative towels (before and after LSCS) and amount of blood in suction unit will be recorded.
* Fluid monitoring will be performed through rate of infusion and urine output. A complete blood count test will be performed 12 hours after delivery.
* Estimated Blood Loss (EBL) will be evaluated as follows:
* The number of operative towels used.
* The difference of weight of operative towels (before and after cs) plus the amount of blood in suction unit (we will calculate 1 gram of weight difference equal to 1 ml blood loss).
* EBL calculation according to the formula which is EBL equals EBV times Preoperative hematocrit minus Postoperative hematocrit divided by Postoperative hematocrit.
* Where EBV is estimated blood volume of the patient in mL (equals weight in kg × 85).
* In Tranexamic Acid group (n=111), the time interval between drug administration and fetal delivery will be recorded.
* All patients will be followed up following the delivery as regard occurrence of primary postpartum hemorrhage (within the first 24 hours), the need for blood transfusion (within the first 24 hours), misoprostol-related side effects (in the first 6 hours) (i.e., shivering, pyrexia >38C0, headache, nausea, vomiting with or without the need for antiemetic drugs), carbetocin - related side effects (i.e., nausea, vomiting, flushing, dizziness, syncope) and the occurrence of thromboembolic events (within one week of delivery).
* The EBL will be compared among the four groups together with occurrence of the above-mentioned drugs side effects.

ELIGIBILITY:
Inclusion Criteria:

* 2. Pregnant women candidate for LSCS. 3. Age: 20-40 years old. 4. Full term pregnancies (> 37 weeks confirmed by the 1st day of the LMP or 1st trimesteric ultrasound scan).

  5. Singleton pregnancies. 6. One or more of the following criteria to be considered as high-risk case for PPH (RCOG, 2016):
  1. Maternal Anemia (hemoglobin < 10 g%).
  2. Known placenta previa.
  3. Proven or suspected case of placental abruption.
  4. Preeclampsia or gestational hypertension.
  5. Polyhydramnios (DVP > 8cm).
  6. Macrosomia (> 4 Kg)
  7. Previous history of uterine atony or postpartum hemorrhage).
  8. Prolonged labour (>12 hours).

     7. CS under spinal anesthesia.

     Exclusion Criteria:
* 1. Fetal death (IUFD). 2. Fetal anomalies. 3. IUGR (Estimated fetal weight below the 5th centile) 4. Women presenting with an obstetric emergency necessitating immediate surgery (Cord prolapse, severe antepartum hemorrhage, severe fetal distress etc.) 5. More than 2 previous CS procedures. 6. Prolonged procedure (more than 2 hours from skin incision to skin closure). 7. History of prostaglandin, Tranexamic acid or carbetocin allergy. 8. Multifetal pregnancies. 9. Abnormally invasive placenta. 10. Known deep venous thrombosis

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Estimated Blood Loss | 1 year
  To compare the estimated blood loss (EBL) during and after cesarean delivery among the four groups.

SECONDARY OUTCOMES:
Need for additional ecbolics | 1 year
  The Use of additional ecbolics denoting uterine atony (i.e. 10 IU intravenous infusion of oxytocin with 500 ml lactated ringer at a rate of 125 ml/hour and 1mL [0.2 mg] intramuscular ergometrine with or without 600 microgram rectal misoprostol postoperatively)
Excessive blood loss and need for blood transfusion | 1 year
  The occurrence of excessive blood loss (> 1000 mL) together with the need for blood transfusion within the first 24 hours postoperatively.
Side effects | 1 year
  The occurrence of any maternal side effects (among the four groups).

CONTACTS AND LOCATIONS:
Overall Officials: Amr K Rasheed, MsC, Principal Investigator — Assistant Lecturer, Cairo University
Locations (2):
- Egypt (2):
  - kasr elainy hospital (Faculty of Medicine - Cairo University), Cairo
  - Faculty of medicine - Cairo university, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen CY, Su YN, Lin TH, Chang Y, Horng HC, Wang PH, Yeh CC, Chang WH, Huang HY. Carbetocin in prevention of postpartum hemorrhage: Experience in a tertiary medical center of Taiwan. Taiwan J Obstet Gynecol. 2016 Dec;55(6):804-809. doi: 10.1016/j.tjog.2016.07.009. PMID 28040124
- [Result] Prata N, Weidert K. Efficacy of misoprostol for the treatment of postpartum hemorrhage: current knowledge and implications for health care planning. Int J Womens Health. 2016 Jul 29;8:341-9. doi: 10.2147/IJWH.S89315. eCollection 2016. PMID 27536161
- [Result] Della Corte L, Saccone G, Locci M, Carbone L, Raffone A, Giampaolino P, Ciardulli A, Berghella V, Zullo F. Tranexamic acid for treatment of primary postpartum hemorrhage after vaginal delivery: a systematic review and meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2020 Mar;33(5):869-874. doi: 10.1080/14767058.2018.1500544. Epub 2018 Sep 10. PMID 30122082